CLINICAL TRIAL: NCT02400593
Title: An Affective Intervention to Reverse the Biological Residue of Low Childhood SES
Brief Title: Health Experiences & Early Life Disadvantages
Acronym: HEELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Barbara L. Fredrickson, PhD, Kenan Distinguished Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-1938; R01AG048811 (NIH)
Record Dates: First submitted 2015-03-23; First posted 2015-03-27 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Early Life Adversity; Chronic Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovingkindness (Experimental): A six-week formal meditation workshop for 1 hour per week.
  Interventions: Behavioral: Meditation Workshop
- Mindfulness (Placebo Comparator): A six-week formal meditation workshop for 1 hour per week.
  Interventions: Behavioral: Meditation Workshop

INTERVENTIONS:
Behavioral: Meditation Workshop — Six weeks of formal instruction in Lovingkindness or Mindfulness meditation.

SUMMARY:
Growing up in a low-income household has been shown to increase risk for, and susceptibility to many illnesses.The purpose of the study is to test an affective intervention for reversing biological risk factors, as related to childhood adversity, in midlife.

Participants will be asked to make two lab visits; attend six weekly, 1-hour meditation classes; as well as complete brief online daily surveys for 11 weeks, five biweekly surveys, and two 30-minute surveys prior to each lab visit. During the lab visits, participants will have their psychophysiology monitored for heart rate, blood pressure, respiration, and pulse. Participants will also have their blood drawn.

All surveys and questionnaires inquire about participants' current demographics, family history, perceptions about life and well-being, physical health, and monetary choices.

ELIGIBILITY:
Inclusion Criteria:

* fluent in written and spoken English
* have daily access to internet and a computer

Exclusion Criteria:

* engaged in regular meditation practice, either recently or in the past
* previously participated in a meditation study
* have allergies to adhesive materials (includes latex)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in meditation time (Self-reported meditation time recorded daily) | Weeks 3, 4, 5, 6, 7, 8, 9 ,10, 11, 12
  Self-reported meditation time recorded daily.

SECONDARY OUTCOMES:
Leukocyte basal gene expression (evaluated through blood samples) | Week 0, Week 12
  Gene expression evaluated through blood samples.
Levels of mistrust (Self-report questionnaire measure of hostility using 9-item Cooke-Medley scale) | Week 0, Week 12
  Self-report questionnaire measure of hostility using 9-item Cooke-Medley scale.
Temporal Discounting (Monetary choice questionnaire to assess impulsive decision-making) | Week 0, Week 12
  Monetary choice questionnaire to assess impulsive decision-making.
Cardiac vagal tone (Respiration and echocardiogram measured with respiration band and 2-lead electrode placement) | Week 0, Week 12
  Respiration and echocardiogram measured with respiration band and 2-lead electrode placement, respectively. Three-minute spontaneous breath followed by five minutes of paced breathing intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Fredrickson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC PEP Lab, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Miller GE, Chen E, Fok AK, Walker H, Lim A, Nicholls EF, Cole S, Kobor MS. Low early-life social class leaves a biological residue manifested by decreased glucocorticoid and increased proinflammatory signaling. Proc Natl Acad Sci U S A. 2009 Aug 25;106(34):14716-21. doi: 10.1073/pnas.0902971106. Epub 2009 Jul 14. PMID 19617551
- [Background] Cohen S, Doyle WJ, Turner RB, Alper CM, Skoner DP. Childhood socioeconomic status and host resistance to infectious illness in adulthood. Psychosom Med. 2004 Jul-Aug;66(4):553-8. doi: 10.1097/01.psy.0000126200.05189.d3. PMID 15272102
- [Background] Miller GE, Chen E, Parker KJ. Psychological stress in childhood and susceptibility to the chronic diseases of aging: moving toward a model of behavioral and biological mechanisms. Psychol Bull. 2011 Nov;137(6):959-97. doi: 10.1037/a0024768. PMID 21787044
- [Background] Cole SW, Hawkley LC, Arevalo JM, Cacioppo JT. Transcript origin analysis identifies antigen-presenting cells as primary targets of socially regulated gene expression in leukocytes. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3080-5. doi: 10.1073/pnas.1014218108. Epub 2011 Feb 7. PMID 21300872
- [Background] Kok BE, Fredrickson BL. Upward spirals of the heart: autonomic flexibility, as indexed by vagal tone, reciprocally and prospectively predicts positive emotions and social connectedness. Biol Psychol. 2010 Dec;85(3):432-6. doi: 10.1016/j.biopsycho.2010.09.005. Epub 2010 Sep 22. PMID 20851735
- [Derived] West TN, Zhou J, Brantley MM, Kim SL, Brantley J, Salzberg S, Cole SW, Fredrickson BL. Effect of Mindfulness Versus Loving-kindness Training on Leukocyte Gene Expression in Midlife Adults Raised in Low-Socioeconomic Status Households. Mindfulness (N Y). 2022 May;13(5):1185-1196. doi: 10.1007/s12671-022-01857-z. Epub 2022 Mar 16. PMID 36278141